CLINICAL TRIAL: NCT02651896
Title: Hypofractionated Intensity Modulated and Image Guided Radiotherapy for Localized Prostate Cancer: a Prospective Cohort.
Brief Title: Hypofractionated Intensity Modulated and Image Guided Radiotherapy for Localized Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Rafael Gadia, Head of Radiation Oncology - Hospital Sírio Libanês - Unidade Brasília, Hospital Sirio-Libanes
Other Study IDs: HSL 2015-64
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HypoIGRT: 1. Low Risk (T1-T2a, Gleason score 6, and PSA < 10 ng/mL)
  2. Intermediate Risk (T1-T2c, Gleason 7, and PSA 10-20 ng/mL)
  3. High Risk (T3 - 4 , Gleason 8-10, and/or PSA > 20 ng/mL) Neoadjuvant hormone therapy is allowed on groups 2 and 3
  Interventions: Radiation: HypoIGRT

INTERVENTIONS:
Radiation: HypoIGRT — Hypofractionated intensity modulated and image guided radiotherapy 60 Gy in 20 fractions over four weeks for the prostate gland to all groups.
  For intermediate and high risk group: seminal vesicle will be included: 48 Gy in 20 fractions over 4 weeks (proximal third to half on physicians description).
  Image guidance with cone beam CT will be mandatory before every treatment fraction.

SUMMARY:
Hypofractionated intensity modulated and image guided radiotherapy (HypoIGRT) with fewer high-fraction-size treatments would be beneficial for prostate cancer because it would deliver a larger biological-equivalent dose to the tumor than would conventional treatment in 1.8-2.0 Gy fractions, while maintaining a similar or lower incidence of late normal tissue reactions. Thus, the investigators aim to assess the hypothesis that HypoIGRT treatment for localized prostate cancer will improve the therapeutic ratio by either:

1. Reducing normal tissue, mainly genitourinary and gastrointestinal, toxicity and / or
2. Improving tumour control, mainly freedom from biochemical failure survival.

DETAILED DESCRIPTION:
The investigator chose to study a HypoIGRT regimen, in participants with prostate adenocarcinoma, tumor which is considered to present a low α / β, and therefore benefit from this approach.

Primary Outcome Measures:

1. Acute and late radiation induced toxicities.

Secondary Outcome Measures:

1. Freedom from prostate cancer recurrence - freedom from biochemical failure survival;
2. Cause specific and overall survival
3. Aspects of quality of life and health economics

Study Design:

Allocation: Prospective allocation Endpoint Classification: Feasibility Study (Toxicity assessment) Intervention Model: Single Assignment Masking: Open Label Primary Purpose: Treatment

Eligibility

Ages Eligible for Study: 18 Years and older Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Study Population:

Men with localized histologically confirmed T1B-T4 N0 and M0 prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, previously untreated locally confined adenocarcinoma of the prostate
2. Patients older than 18 years old
3. Patients who accept to perform follow up in the radiation oncology department
4. Performance Status ≥ 70
5. Written informed consent

Exclusion Criteria:

1. Prior pelvic radiotherapy, radical prostatectomy, brachytherapy, cryotherapy or other local treatment
2. Presenting with positive pelvic lymph nodes or metastatic at the diagnosis (M1)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with localized histologically confirmed T1B-T4 N0 and M0 prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2015-12-20 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall Acute Gastrointestinal Toxicity - According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. | During and up to 90 days after treatment ends (acute event)
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0 - toxicity will be graduated in a scale from 0 - 5
Overall Acute Genitourinary Toxicity - According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. | During and up to 90 days after treatment ends (acute event)
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0 - toxicity will be graduated in a scale from 0 - 5
Overall Late Gastrointestinal Toxicity - According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. | After 90 days up to 24 months from treatment (late event)
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0 - toxicity will be graduated in a scale from 0 - 5.
Overall Late Genitourinary Toxicity - According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. | After 90 days up to 24 months from treatment (late event)
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0 - toxicity will be graduated in a scale from 0 - 5.

SECONDARY OUTCOMES:
Freedom from biochemical failure survival | 12 and 24 months
  Prostate-Specific Antigen (PSA) values
Overall Survival | 12 and 24 months
  Defined as the percentage of participant on treatment group who are alive at 12 and 24 months after the start of treatment.
Cause specific Survival | 12 and 24 months
  Defined as the cancer survival in the absence of other causes of death at 12 and 24 months after the start of treatment.
Quality of life | 12 and 24 months
  The Expanded Prostate Cancer Index Composite (EPIC) - Brazilian Portuguese version.
  will be applied to assess urinary, bowel and sexual functions.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Reis, MD, PhD, Study Director — Hospital Sírio-Libanes - Ensino e Pesquisa
Locations (2):
- Brazil (2):
  - Hospital Sírio-Libanes, Brasília, Federal District
  - Hospital Sírio-Libanes, São Paulo, São Paulo

REFERENCES:
- [Background] Chang P, Szymanski KM, Dunn RL, Chipman JJ, Litwin MS, Nguyen PL, Sweeney CJ, Cook R, Wagner AA, DeWolf WC, Bubley GJ, Funches R, Aronovitz JA, Wei JT, Sanda MG. Expanded prostate cancer index composite for clinical practice: development and validation of a practical health related quality of life instrument for use in the routine clinical care of patients with prostate cancer. J Urol. 2011 Sep;186(3):865-72. doi: 10.1016/j.juro.2011.04.085. Epub 2011 Jul 23. PMID 21788038
- [Background] Leborgne F, Fowler J. Late outcomes following hypofractionated conformal radiotherapy vs. standard fractionation for localized prostate cancer: a nonrandomized contemporary comparison. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1441-6. doi: 10.1016/j.ijrobp.2008.10.087. Epub 2009 Apr 22. PMID 19395194
- [Background] Moraes FY, Siqueira GM, Abreu CE, da Silva JL, Gadia R. Hypofractioned radiotherapy in prostate cancer: is it the next step? Expert Rev Anticancer Ther. 2014 Nov;14(11):1271-6. doi: 10.1586/14737140.2014.972380. PMID 25367322
- [Background] Dearnaley D, Syndikus I, Sumo G, Bidmead M, Bloomfield D, Clark C, Gao A, Hassan S, Horwich A, Huddart R, Khoo V, Kirkbride P, Mayles H, Mayles P, Naismith O, Parker C, Patterson H, Russell M, Scrase C, South C, Staffurth J, Hall E. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: preliminary safety results from the CHHiP randomised controlled trial. Lancet Oncol. 2012 Jan;13(1):43-54. doi: 10.1016/S1470-2045(11)70293-5. Epub 2011 Dec 12. PMID 22169269
- See also: Protocol team hospital website. — http://hsl.org.br